CLINICAL TRIAL: NCT05952154
Title: Minimally Invasive Transapical Beating-Heart Septal Myectomy in Patients With Nonobstructive Hypertrophic Cardiomyopathy
Brief Title: Transapical Beating-Heart Septal Myectomy in Patients With Symptomatic Nonobstructive Hypertrophic Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiang Wei (Other)
Responsible Party: Sponsor-Investigator, Xiang Wei, Professor and Director, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-S015
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Nonobstructive Hypertrophic Cardiomyopathy
Keywords: Nonobstructive Hypertrophic Cardiomyopathy; Septal Myectomy; Mitral Regurgitation; Transapical; Off-pump; Minimally invasive
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Experimental Group: Beating-heart myectomy device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nonbstructive Hypertrophic Cardiomyopathy (Experimental): Transapical beating-heart septal myectomy for the patient with nonobstructive hypertrophic cardiomyopathy and Heart Failure.
  Interventions: Procedure: Transapical beating-heart septal myectomy

INTERVENTIONS:
Procedure: Transapical beating-heart septal myectomy — We have invented a beating-heart myectomy device.Through a minimally invasive intercostal incision, septal myectomy could be accomplished via a transapical access in the beating heart using the device. The whole process of resection is monitored, navigated, and evaluated by real-time transesophageal and transthoracic echocardiography. Left ventricular end-diastolic volume and the grade of mitral regurgitation are evaluated each time after resection. Multiple resections are performed to tailor the muscular resection for sufficient enlargement of left ventricular end-diastolic volume and improvement of mitral regurgitation, while preventing iatrogenic injuries.
  Other Names: Minimally invasive transapical septal myectomy in the beating hearts

SUMMARY:
The primary purpose of this study is to evaluate the feasibility, the safety and the efficacy of the transapical beating-heart septal myectomy for the treatment of nonobstructive hypertrophic cardiomyopathy. This is a prospective, single-arm, single-center study.

DETAILED DESCRIPTION:
Medical therapy is first recommended for patients with nonobstructive hypertrophic cardiomyopathy administrated at onset of heart failure symptoms. As the disease progresses, patients with global ejection fraction < 50% should be evaluated with respect to eligibility and motivation for heart transplant. However, for those with preserved ejection fraction and drug-refractory heart failure symptoms, there is still no optimal therapy. Some patients with increased left atrial volume and/or diastolic dysfunction can be recognized as a result of excessive myocardial hypertrophy, and the septal resection for these patients may be beneficial. However, conventional septal myectomy is hindered by the demanding expertise that is needed to sufficient resection of hypertrophied septal myocardium while guarantee safety. To increase the visualization and minimize the surgical injury of conventional septal myectomy, we have invented a novel beating-heart myectomy device. Through a mini-thoractomy, septal myectomy could be accomplished via a transapical access in the beating heart using the beating-heart myectomy device. The whole process of resection is monitored, navigated, and evaluated by real-time transesophageal and transthoracic echocardiography. Left ventricular morphology and hemodynamics are evaluated each time after resection. Multiple resections are performed to tailor sufficient enlargement of left ventricular end-diastolic volume and improvement of mitral regurgitation, while preventing iatrogenic injuries. After transapical beating-heart septal myectomy, patients are scheduled to be seen for follow-up visits at discharge (about 7 days post operation) and 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose maximal ventricular septal wall thickness ≥ 15 mm.
2. Patients with heart function of New York Heart Association ≥ class II.
3. Patients with drug-refractory symptoms or intolerable to pharmaceutical therapies.
4. Patients who was informed the nature of the clinical trial, consented to participate in all of the activities of the clinical trial, and signed the informed consent form

Exclusion Criteria:

1. Patients who were pregnant.
2. Patients who had concomitant diseases such as intrinsic valvular disease or coronary artery disease that needed open-heart surgery.
3. Patients who had severe heart failure with left ventricle ejection fraction < 40%.
4. Patients whose estimated life expectancy < 12 m.
5. Patient who were non-compliant.
6. Patients under circumstances which were considered not suitable or prohibitive for participating the clinical trial at the discretion of the attending medical team and the researchers.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 3 months
  Death from any cause during the observation period.
Procedural success | 3 months
  A reduction of ≥1 New York Heart Association (NYHA) class and a decrease of ≥ 20% of left atrial volume

SECONDARY OUTCOMES:
Device success | 1 day
  Successful accession, delivery, and retrieval of the resection device, successful resection of the septal myocardium, mitral regurgitation (MR) ≤ grade 2+ during operation after resection, and free from conversion to midline thoracotomy during operation.
Septal thickness | 7 days and 3 months
  Basal and mid septal thickness as measured by echocardiography.
Left ventricle mass | 7 days and 3 months
  Left ventricle mass index (the ratio of left ventricle mass to body weight) as measured by cardiac magnetic resonance.
Left atrial volume | 7 days and 3 months
  The left atria volume as measured by echocardiography.
Major adverse cardiovascular and cerebral events | 3 months
  In-hospital mortality, atrioventricular block that need permanent pacemaker implantation, sternotomy conversion, iatrogenic ventricular septal perforation, iatrogenic valvular injury, imaging examination-validated cerebral complications.
New York Heart Association class | 7 days and 3 months
  New York Heart Association class, including grade I, grade II, grade III, grade IV. A higher grade means worse heart function.
6-minute walking test | 3 months
  6-minute walking test. A longer distance means better heart function.
Heart function-associated quality of life | 7 days and 3 months
  Score of the Kansas City Cardiomyopathy Questionnaire. A higher score means better heart function.
Evaluation of the mitral valve | 7 days and 3 months
  Grade of mitral regurgitation and systolic anterior motion as measured by echocardiography.
Left ventricular outflow tract diameter | 7 days and 3 months
  Left ventricular outflow tract diameter as measured by echocardiography.
Left ventricular end-diastolic volume | 3 months
  Left ventricular end-diastolic volume as measured by cardiac magnetic resonance.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
All of the conclusive participant data, after removing the individual information of privacy, will be uploaded as supporting information when publishing the current study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the current study is published.
Access Criteria: All readers who were interested in the current study.

REFERENCES:
- [Background] Fang J, Wang R, Liu H, Su Y, Chen J, Han X, Wei Y, Chen Y, Cheng L, Wei X. Transapical septal myectomy in the beating heart via a minimally invasive approach: a feasibility study in swine. Interact Cardiovasc Thorac Surg. 2020 Feb 1;30(2):303-311. doi: 10.1093/icvts/ivz249. PMID 31642911